CLINICAL TRIAL: NCT04723888
Title: The Intervention Effect Of Alpha-Ketoglutarate On Abdominal Aortic Aneurysm Progression and Rupture: A Prospective, Randomized Parallel Controlled Study Based On Large Cohorts
Brief Title: Alpha-Ketoglutarate and Abdominal Aortic Aneurysm Progression and Rupture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jun Pu, Director of Cardiovascular Medicine, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AKG Intervention study
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Patients With an Abdominal Aortic Aneurysm of 39-49 mm in Diameter
Keywords: cohort study
MeSH Terms: interventions — Ketoglutaric Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alpha-ketoglutarate Group (Experimental): Take alpha-ketoglutarate supplements, alpha-ketoglutarate 300mg/d mixed with food or drink, for 1 years
  Interventions: Dietary Supplement: alpha-ketoglutarate
- Normal Control Group (No Intervention): Don't take alpha-ketoglutarate supplements

INTERVENTIONS:
Dietary Supplement: alpha-ketoglutarate — alpha-ketoglutarate supplements
  Arms: alpha-ketoglutarate Group

SUMMARY:
The objective of this project is to define whether nutritional supplement (oral administration with alpha-ketoglutarate) capable of filling-up the citric acid cycle (anaplerotic therapy) can improve outcomes in patients with an abdominal aortic aneurysm of 39-49 mm in diameter on ultrasound imaging. Alpha-ketoglutarate is commonly used as a nutritional supplement specially by athletes to increase muscle strength. They can be mixed with formula or other foods. Subjects will be followed for up to 5 years.

DETAILED DESCRIPTION:
Abdominal aortic aneurysm (AAA) is an age-related disease that characterized by permanent regional dilation of the abdominal aortae, which results in catastrophic event of rupture and sudden death. Currently, no effective drug to limit the progression or reduce the risk of rupture has been developed.

Metabolic pathways, including glucose metabolism, lipid metabolism, and amino acid metabolism, have indispensable roles in normal and dysfunctional vasculature. The Krebs cycle is responsible for obtaining energy from food in the form of ATP, and ATP is essential for muscle contraction and correct functioning of all organs. Besides, tight control of mitochondrial functions is critical for maintaining metabolism balance.

As an important metabolite in Krebs cycle, alpha-ketoglutarate not only improved energy metabolism, but also extended lifespan and reduced morbidity in aging mice. It is widely used in the market as a nutritional supplement specially by athletes to increase muscle strength. Until now, no obvious toxic and side effects to the body was observed. Given the high bioavailability, we propose that dietary supplementation with alpha-ketoglutarate can improve the outcome in patients with an abdominal aortic aneurysm of 39-49 mm in diameter.

Therefore, the project team intends to establish the abdominal aortic aneurysm rupture risk prediction model in the elderly cohort in the early stage, and randomize groups in patients with an abdominal aortic aneurysm of 39-49 mm in diameter based on whether or not to supplement alpha-ketoglutarate. There are two cohorts: the alpha-ketoglutarate intervention cohort and the parallel control cohort. By observing the efficacy in terms of change in aortic diameter and abdominal aortic aneurysm rupture incidence in the two groups during the follow-up period, it provides evidence-based medical evidence for the future clinical application of alpha-ketoglutarate.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of an infrarenal AAA with a maximum diameter of 39-49 mm;
2. Han nationality;
3. Between 50 years or more, no gender limit;
4. No mental illness;
5. No history of supplement allergy or supplement allergy;
6. Subjects voluntarily participate in this study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Exclusion Criteria:

1. Previous infrarenal aortic surgery;
2. Planned major surgery;
3. Known aortic dissection;
4. Have received any other clinical trial treatment within 1 year;
5. Systemic treatment with corticosteroids or other systemic immunomodulatory therapy;
6. Severe infections, including but not limited to infections requiring hospitalization, bacteremia, severe pneumonia, etc.;
7. Known or suspected inherited connective tissue disorder;
8. Calculated creatinine clearance of less than 30 ml/min;
9. Known significant liver disease;
10. Known human immunodeficiency virus infection at the time of screening；
11. Serious concomitant illness associated with life expectancy of less than 2 years；
12. Any other significant and unstable condition that could limit compliance with the trial protocol.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in aortic diameter | 1 year
  Measure the aortic diameter by ultrasound imaging from leading edge adventitia at the anterior wall to leading edge adventitia at the posterior wall.

SECONDARY OUTCOMES:
Rates of AAA repair/rupture | 1 year
  Calculate the incidence of AAA repair/rupture
Rates of mortality | 1 year
  Calculate the mortality due to AAA rupture
Changes level of plasma biomarker | 1 year
  Measure plasma levels of tryptase

CONTACTS AND LOCATIONS:
Overall Officials: Jun Pu, Principal Investigator — RenJi Hospital
Locations (1):
- Cardiology, Ren Ji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No